CLINICAL TRIAL: NCT01210846
Title: An Open-Label Cardiac Safety Study of Tivozanib to Evaluate the Electrocardiogram and Pharmacokinetic-Electrocardiogram Dynamics in Subjects With Advanced Solid Tumors
Brief Title: A Cardiac Safety Study of Tivozanib to Evaluate the Electrocardiogram and Pharmacokinetic-Electrocardiogram Dynamics in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AV-951-10-112
Record Dates: First submitted 2010-09-27; First posted 2010-09-29 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Advanced Solid Tumors
Keywords: AV-951; tivozanib; QTc; advanced solid tumors; pharmacokinetics
MeSH Terms: interventions — tivozanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tivozanib (Experimental)
  Interventions: Drug: tivozanib

INTERVENTIONS:
Drug: tivozanib — 1 x 1.5 mg capsule of tivozanib orally once daily for 21 days

SUMMARY:
The purpose of this study is to obtain QTc data, to assess the effects of tivozanib on ECG morphology, and to determine the pharmacokinetic pharmacodynamic (PK-PD) relationship between any observed changes in cardiac repolarization (defined by QTcF duration) and the serum concentration of tivozanib.

DETAILED DESCRIPTION:
Tivozanib is a novel and potent pan-vascular endothelial growth factor (VEGF) receptor (VEGFR) tyrosine kinase inhibitor with potent activity against all 3 VEGFRs (VEGFR-1, -2, and -3). In nonclinical models and studies performed in humans, tivozanib has shown strong antiangiogenesis and antitumor activity.

This study is an open-label, non-randomized, exploratory single-arm trial evaluating the ECG and pharmacokinetic (PK)-ECG relationship, if any, of tivozanib in subjects with advanced solid tumors.

The purpose of this study is to evaluate the ECG intervals and morphology following treatment with tivozanib in subjects with advanced solid tumors and to determine the relationship, if any, of the change in QTc duration with serum concentration of tivozanib over time in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria

* Males or females, ≥18 years of age;
* Diagnosis of an advanced solid tumor malignancy with histological or cytological evidence;
* Advanced malignancy, metastatic or unresectable, that has recurred or progressed following standard therapy or failed standard therapy; or for which no standard therapy currently exists; or for which subject is not a candidate, or is unwilling to undergo standard therapy;
* Tumor is not currently amenable to curative surgical intervention;
* Recovery from the effects of any prior surgery, radiotherapy, or systemic antineoplastic therapy;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, and life expectancy ≥ 3 months;
* Well controlled thyroid function, in the opinion of the Investigator;
* Able to comprehend and willing to sign an Informed Consent Form (ICF) and able to adhere to dose and visit schedule.

Exclusion Criteria

- Women who are breast-feeding, pregnant, or intend to become pregnant;

* Primary central nervous system (CNS) malignancies or CNS metastases; subjects with previously treated brain metastasis will be allowed if the brain metastasis have been stable without steroid treatment for at least 3 months following prior treatment (radiotherapy or surgery);
* Clinically significant cardiac disease (New York Heart Association class > 2) including unstable angina, acute myocardial infarction within 6 months of Day 1, congestive heart failure, or arrhythmia requiring therapy, with the exception of extra systoles or minor conduction abnormalities, per Investigator judgment;
* Uncontrolled hypertension: systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg on 2 or more antihypertensive medications, documented on 2 consecutive measurements taken at least 24 hours apart;
* Baseline ECG, QTcF > 480 ms. If the screening QTcF is > 480 ms, this may be repeated once and if the QTcF is ≤ 480 ms the subject can be enrolled;
* Any of the following hematologic abnormalities:

  • hemoglobin < 9.0 g/dL;

  • Absolute neutrophil count < 1500 per mm3;
  * platelet count < 100,000 per mm3;
  * INR > 1.5 x upper limit of normal (ULN);
* Any of the following serum chemistry or urine abnormalities:

  • total bilirubin > 1.5 × ULN (or > 2.5 × ULN for subjects with Gilbert's syndrome);
  * AST or ALT > 2.5 × ULN (or > 5 × ULN for subjects with liver metastasis);
  * alkaline phosphatase > 2.5 × ULN (or > 5 × ULN for subjects with liver or bone metastasis);
  * creatinine > 2.0 × ULN;
  * proteinuria > 3+ by urinalysis;
* Non healing wound, bone fracture, or skin ulcer;
* Active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, or other gastrointestinal condition with increased risk of perforation; history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 4 weeks prior to administration of first dose of study drug;
* Serious/active infection or infection requiring parenteral antibiotics or antifungal therapy;
* Inadequate recovery from any prior surgical procedure or major surgical procedure within 4 weeks prior to administration of first dose of study drug;
* Significant thromboembolic or vascular disorders or surgery within 6 months prior to administration of first dose of study drug, including but not limited to:

  • deep vein thrombosis;

  • pulmonary embolism;

  • cerebrovascular accident or transient ischemic attack;

  • peripheral arterial ischemia > Grade 2;

  • coronary or peripheral artery bypass graft;
* Significant bleeding disorders within 6 months prior to administration of first dose of study drug, including but not limited to:

  • hematemesis, hematochezia, melena or other gastrointestinal bleeding ≥ Grade 2;
  * hemoptysis or other pulmonary bleeding ≥ Grade 2;
  * hematuria or other genitourinary bleeding ≥ Grade 2;
* Currently active second primary malignancy, including hematologic malignancies (leukemia, lymphoma, multiple myeloma, etc), other than non melanoma skin cancers, non-metastatic prostate cancer, in situ cervical cancer and ductal or lobular carcinoma in situ of the breast. Subjects are not considered to have a currently active malignancy if they have completed anti-cancer therapy and have been disease free for >2 years;
* History of genetic or acquired immune suppression disease such as human immunodeficiency virus (HIV), subjects on immune suppressive therapy for organ transplant;
* Life-threatening illness or organ system dysfunction compromising safety evaluation;
* Inability to swallow pills, malabsorption syndrome or gastrointestinal disease that severely affects the absorption of tivozanib, major resection of the stomach or small bowel, or gastric bypass procedure;
* Psychiatric disorder or altered mental status precluding informed consent or necessary testing;
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator;
* Use of Seville orange- or grapefruit-containing foods or beverages within 72 hours prior to Day 1;
* Poor venous access;
* Any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study;
* Sexually active male and pre-menopausal female subjects (and their partners) unless they agree to use adequate contraceptive measures, while on study and for 30 days after the last dose of study drug. All fertile male and female subjects (and their partners) must agree to use a highly effective method of contraception. Highly effective birth control includes (a) IUD plus one barrier method; or (b) two barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm). Note: Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are not considered effective for this study.

Drugs and Other Treatments to be Excluded

Prohibited 4 weeks prior to first dose and for the duration of the study:

- Chemotherapy, biological therapy (including cytokines, signal transduction inhibitors, monoclonal antibodies), immunotherapy, experimental therapy or any other therapy for treatment of advanced solid tumors;

- Systemic hormonal therapy, with the exception of: i. hormonal therapy for appetite stimulation or contraception; ii. nasal, ophthalmic, inhaled and topical steroid preparations; iii. androgen suppression therapy for non-metastatic prostate carcinoma; iv. hormone replacement therapy for conditions such as adrenal insufficiency, hypothyroidism, etc.; v. low-dose maintenance steroid therapy (equivalent of prednisone ≤ 10 mg/day) for other conditions;

Prohibited 3 weeks prior to first dose and for the duration of the study:

- Treatment with radiotherapy (limited radiotherapy involving ≤ 25% of bone marrow may be allowed for palliative purposes after consultation with the medical monitor, treatment with study drug must be stopped during radiotherapy);

Prohibited 2 weeks prior to first dose and for the duration of the study:

* Herbal preparations/supplements/topical applications (except for daily multivitamin/mineral supplement not containing herbal components);
* Treatment with CYP3A4 inducers or inhibitors (see Appendix C for examples);

Prohibited 1 week prior to first dose and for the duration of the study:

- Treatment with full dose oral anticoagulants such as warfarin, acenocoumarol, fenprocoumon, or similar agents. If previously receiving these types of agents, a minimum washout of 1 week and documented PT of < 1.5 × ULN will be required prior to start of therapy. Full dose anticoagulation with low molecular weight heparin or unfractionated heparin administered subcutaneously is allowed. Low dose oral anticoagulation (eg, 1-2 mg/day warfarin) is allowed provided PT remains < 1.5 × ULN during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QTcF | 22 days

SECONDARY OUTCOMES:
Change from baseline in QTc with Bazett correction method (QTcB) | 22 days
Change from baseline in heart rate (HR) | 22 days
Change from baseline in PR interval | 22 days
Change from baseline in QRS interval | 22 days
Change from baseline in Uncorrected QT interval | 22 days
Change from baseline in ECG morphological patterns | 22 days
Correlation between the QTcF change from baseline and serum concentrations of tivozanib | 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Vargo, MD, Study Director — AVEO Pharmaceuticals, Inc.
Locations (8):
- United States (8):
  - TGEN Clinical Research Service at Scottsdale Healthcare, Scottsdale, Arizona
  - Florida Cancer Specialists, Fort Myers, Florida
  - Horizon Oncology Research, Inc., Lafayette, Indiana
  - Jayne Gurtler MD, Laura Brinz MD, Angelo Russo MD and Janet Burroff MD APMC, Metairie, Louisiana
  - Associates in Oncology/Hematology, Rockville, Maryland
  - Oklahoma University Cancer Institute (OUCI), Oklahoma City, Oklahoma
  - Tennessee Onocology, Nashville, Tennessee
  - Multicare Research Institute/Tacoma General Hospital, Tacoma, Washington